CLINICAL TRIAL: NCT05387642
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Trial to Explore the Safety, Tolerability, Pharmacokinetics, and Efficacy of PRAX-114 in the Treatment of Adults With Essential Tremor
Brief Title: A Clinical Trial of PRAX-114 in Participants With Essential Tremor
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor no longer pursuing indication.
Sponsor: Praxis Precision Medicines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRAX-114-231
Record Dates: First submitted 2022-05-13; First posted 2022-05-24 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Essential Tremor
Keywords: Essential Tremor; Tremor; GABAA; GABAA receptor; GABAA PAM; Movement Disorders; Central Nervous System Diseases
MeSH Terms: conditions — Essential Tremor; Tremor; Movement Disorders; Central Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Double-blind Sequence 1 (Experimental): Double-blind treatment sequence of 10 mg, 20 mg, and placebo in the morning
  Interventions: Drug: 10 mg PRAX-114, 20 mg PRAX-114, and Placebo
- Double-blind Sequence 2 (Experimental): Double-blind treatment sequence of 20 mg, placebo, and 10 mg in the morning
  Interventions: Drug: 10 mg PRAX-114, 20 mg PRAX-114, and Placebo
- Double-blind Sequence 3 (Experimental): Double-blind treatment sequence of placebo, 10 mg, and 20 mg in the morning
  Interventions: Drug: 10 mg PRAX-114, 20 mg PRAX-114, and Placebo
- Open-label Period PRAX-114 (Experimental): Open-label extension period - 10 mg or 20 mg PRAX-114 once daily in the morning for 28 days
  Interventions: Drug: 10 mg PRAX-114 or 20 mg PRAX-114

INTERVENTIONS:
Drug: 10 mg PRAX-114, 20 mg PRAX-114, and Placebo — Single dose with a washout period between doses
  Arms: Double-blind Sequence 1; Double-blind Sequence 2; Double-blind Sequence 3
Drug: 10 mg PRAX-114 or 20 mg PRAX-114 — Once daily oral treatment for 28 days
  Arms: Open-label Period PRAX-114

SUMMARY:
This is a 2-part clinical trial to evaluate the safety, tolerability, pharmacokinetics, and efficacy of PRAX-114 in participants with essential tremor (ET). Part A is a randomized, double-blind, placebo-controlled, three-period, three-sequence, crossover design where participants will receive a single dose of 10 mg PRAX-114, 20 mg PRAX-114, and matching placebo. Part B is an open-label design where participants from Part A, after washout and confirmation of eligibility may elect to participate in Part B where all participants will receive 10 mg once every morning (QAM) for the first 14 days. Based on investigator judgement of the safety and tolerability, the dose for Days 15 to 28 could be increased to 20 mg QAM.

ELIGIBILITY:
Inclusion Criteria:

1. Has a clinical diagnosis of moderate to severe ET, including, a) tremor syndrome of bilateral upper limb action tremor, b) symptoms for at least 3 years in duration, c) with or without tremor in other locations (eg, head, voice, or lower limbs), d) if the symptoms and signs are judged by the investigator to be due to the diagnosis of ET, it is acceptable for them to also have one or more of the following ET plus signs: i) mild dystonic posturing, ii) mild rest tremor in the setting of advanced ET and in the absence of other features of Parkinsonism, iii) intention tremor, iv) mild increase in tandem gait difficulty.
2. Has a TETRAS upper limb score (ie, sum of bilateral upper limb items 4a, 4b, and 4c) of ≥10 as rated by the Investigator at Screening and Baseline. (Exception for Part B only: Tremor severity can fluctuate, and it may be that a participant who met TETRAS upper limb criteria at Screening and Day 1 for Part A no longer meets the tremor severity inclusion criterion above at Screening or on Day 1 of Part B. If all the other eligibility criteria are still met such a participant would still be eligible for inclusion in Part B.)
3. If receiving primidone or topiramate for ET, is willing and able to complete discontinuation no later than 14 days prior to Day 1 of Part A. If currently receiving any other medication for ET, is on a stable dose of any of these other medications for ET for 28 days prior to Screening and is willing to maintain stable doses throughout the clinical trial.
4. Has a body mass index (BMI) between 18 and 40 kg/m2, inclusive.

Exclusion Criteria:

1. Has a history or clinical evidence of other medical, neurological, or psychiatric condition that may explain or cause tremor, including but not limited to Parkinson's disease, Huntington's disease, Alzheimer's disease, cerebellar disease (including spinocerebellar ataxias), primary dystonia, Fragile X Tremor/Ataxia syndrome or family history of Fragile X syndrome, traumatic brain injury, psychogenic tremor, alcohol or benzodiazepine abuse or withdrawal, multiple sclerosis, polyneuropathy, and endocrine states such as hyperthyroidism or unstable treatment of hypothyroidism or medication, food, or supplement induced movement disorders (eg, tremor related to beta agonists or caffeine), or other medical, neurological, or psychiatric conditions that may explain or cause tremor.
2. Has trauma to the nervous system within 3 months preceding the onset of tremor.
3. Has had prior magnetic resonance-guided focused ultrasound or surgical intervention for ET such as deep brain stimulation or thalamotomy.
4. Has had botulinum toxin injection for ET in the 6 months prior to Screening.
5. Is using the Cala trio health device for ET in the last 14 days prior to Baseline and throughout the study.
6. Is unwilling or unable to refrain from episodic use of medication(s)/substance(s) that might interfere with the evaluation of tremor during the trial. Stable use of medication(s)/substance(s) that might impact tremor, including caffeine and beta-agonist bronchodilators, is allowed so long as the tremor is judged by the Investigator to be primarily due to the participant's ET diagnosis.
7. Is unwilling or unable to refrain from use of any sleep aids (eg, eszopiclone, zaleplon and zolpidem) or anxiolytics that are known to be mediated by GABAergic mechanisms (eg, benzodiazepines) within 24 hours prior to any clinic visit. (Exception: Stable use (at least 28 days prior to Screening) of up to 2 ET non-tremor active, non-GABAergic antidepressants and anxiolytics is allowed during the clinical trial after discussion with the medical monitor and/or sponsor designee.) (Note for Part B only: Participants should avoid using sleep aids and anxiolytics that are known to be mediated by GABAergic mechanisms in Part B.)
8. Is unwilling or unable to refrain from alcohol 24 hours before and during clinical trial visits, or regular consumption of more than 2 standard alcohol-containing beverages per day for males or more than 1 standard alcohol-containing beverages per day for females and are unwilling to reduce consumption to the appropriate level during the Screening period and maintain this level throughout the Intervention and Follow-up Periods.
9. Has a history of substance use disorder consistent with Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria in the opinion of the Investigator.
10. Has a lifetime history of seizures, including febrile seizures.
11. Is required to take any excluded medication listed in the protocol during the clinical trial. Chronic medication must be stable for at least 4 weeks prior to Screening. Any new non-urgent medications started during the trial and permitted in protocol should be discussed with the Sponsor before initiation, as practicable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Part A: Incidence and severity of Adverse Events (AE) | 12 days
  The incidence and severity of AEs will be reported by preferred term, including any terms related to clinically significant physical examination findings, as well as vital sign measures (changes in body temperature, pulse rate, respiratory rate, blood pressure [systolic and diastolic]), clinical laboratory measures (chemistry, hematology, urinalysis, and coagulation), electrocardiogram parameters (heart rate, PR, QRS, QT, and corrected QT intervals), Stanford Sleepiness Scale, and Columbia-Suicide Severity Rating Scale (C-SSRS) responses.
Part B: Incidence and severity of AEs | 35 days
  The incidence and severity of AEs will be reported by preferred term, including any terms related to clinically significant physical examination findings, as well as vital sign measures (changes in body temperature, pulse rate, respiratory rate, blood pressure [systolic and diastolic]), clinical laboratory measures (chemistry, hematology, urinalysis, and coagulation), electrocardiogram parameters (heart rate, PR, QRS, QT, and corrected QT intervals), and Columbia-Suicide Severity Rating Scale (C-SSRS) responses.

SECONDARY OUTCOMES:
Part A: Change from pre-dose to each post-dose timepoint on the Essential Tremor Rating Assessment Scale (TETRAS) combined upper limb (CUL) score | Day 1, Day 5, and Day 9
  The TETRAS is an essential tremor and activities of daily living rating scale. The full scale has 2 sections, the Performance subscale (PS) and the TETRAS ADL subscale. The TETRAS PS consists of 9 items covering different body regions. TETRAS CUL aggregates the upper limb items from the TETRAS PS including Items 4, 6, 7 and 8. The total score of the 4 items (9 ratings) ranges from 0 to 44 with higher scores indicating greater tremor severity.
Part B: Change from baseline to Day 28 on the TETRAS Activities of Daily Living (ADL) subscale scores | Day 1, Day 28
  The TETRAS ADL subscale consists of 12 items measuring the impact of essential tremor on typical daily activities. These 12 items are rated on a 5-point scale (ranging from 0 to 4). The total score of the 12 items ranges from 0 to 48 with higher scores indicating greater tremor severity.

CONTACTS AND LOCATIONS:
Overall Officials: VP, Clinical Development, Study Director — Praxis Precision Medicines
Locations (3):
- United States (3):
  - Praxis Research Site, Boca Raton, Florida
  - Praxis Research Site, Farmington Hills, Michigan
  - Praxis Research Site, Kirkland, Washington